CLINICAL TRIAL: NCT03762200
Title: A Prospective, Clinical Study Evaluating the Safety and Haemostatic Effectiveness of SURGICEL® Powder, in Mild or Moderate Parenchymal or Soft Tissue Bleeding During General, Gynaecological, Urological, and Cardiothoracic Surgery
Brief Title: SURGICEL® Powder in Controlling Mild or Moderate Parenchymal or Soft Tissue Intraoperative Bleeding in Adult Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIOS-2017-01
Record Dates: First submitted 2018-11-26; First posted 2018-12-03 (Actual); Results first posted 2020-12-22 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Hemorrhage
Keywords: bleeding; broad area oozing bleeding; hemostat; topical hemostatic agents; adjunctive hemostats
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- SURGICEL Powder - Single arm (Other): Single arm clinical trial where all qualified subjects will be treated SURGICEL Powder
  Interventions: Device: SURGICEL Powder

INTERVENTIONS:
Device: SURGICEL Powder — SURGICEL Powder is a topical absorbable hemostatic treatment made of oxidized regenerated cellulose (ORC) - plant material

SUMMARY:
This is a prospective, single arm, multicentre, multispecialty, post market, clinical study evaluating SURGICEL Powder as an adjunct to achieve haemostasis (control bleeding) when conventional methods of control are impractical or ineffective during surgery (open, laparoscopic or thoracoscopic) in adult subjects (18 years or older).

After application of SURGICEL Powder, the Target Bleeding Site (TBS) will be assessed for haemostasis (no detectable bleeding) at 3, 5, and 10 minutes from application and prior to initiation of closure.

All enrolled subjects will be followed post-operatively through discharge and again at 30 days and 6 months post-surgery via phone call or office visit.

DETAILED DESCRIPTION:
This is an open label, prospective, single arm, multicentre, multispecialty, post-marketing clinical study evaluating SURGICEL Powder as an adjunct to achieve haemostasis in the control of capillary, venous, and small arterial haemorrhage when ligation or other conventional methods of control are impractical or ineffective during surgery (open, laparoscopic or thoracoscopic) in adult subjects (18 years or older). Prospective subjects will be informed about the nature of the research, given the informed consent form (ICF) to read, and, if he/she understands the content, will be asked to provide consent by signing the ICF.

Screening and enrolment will continue until at least 100 evaluable subjects from approximately eight (8) investigational sites, with an appropriate mild or moderate Target Bleeding Site (TBS) are included into the study. The TBS will be the only region evaluated for the primary endpoint and all secondary effectiveness endpoints.

All enrolled subjects will be followed post-operatively through discharge, and via phone call or office visit at 30 days (+14 days) post-surgery. In addition, all enrolled subjects will receive a 6-month (+/-30 days) follow-up phone call or office visit to assess the occurrence of any serious adverse event (SAE) requiring surgical intervention and assessed as possibly related or related to the study treatment.

ELIGIBILITY:
Inclusion Criteria:

Pre-operative:

1. Adult subjects ≥ 18 years requiring elective/non-emergent open or laparoscopic general, gynaecological, cardiothoracic, or urological surgical procedures;
2. Subject or authorised representative has signed the approved Informed Consent;
3. Subject(s) whose International Normalised Ratio is <1.5 within 24 hours of surgery.

   Intra-operative:
4. Presence of an appropriate TBS identified intra-operatively by the surgeon;
5. Subject(s) undergoing cardiothoracic surgery with anticoagulation must have anticoagulation reversed prior to TBS identification and treatment.

Exclusion Criteria:

Pre-operative:

1. Female subjects who are pregnant or nursing;
2. Subject on anticoagulation medication (with exception of aspirin) prior to surgery. Washout periods for respective medications must be observed.

   If information is not readily available within the Instructions for Use (IFU), a conservative approach should be taken and intravenous heparin stopped 12 hours prior to surgery and 2 days prior for oral medication;
3. Subject on antiplatelet/P2Y12 inhibitors medication prior to surgery. Platelet recovery times for respective medication must be observed. If information is not readily available within the IFU, a conservative approach should be taken and medication stopped 5 days prior to surgery.
4. Subject is currently participating or plans to participate in any other investigational device or drug without prior approval from the Sponsor;
5. Subjects who are known, current alcohol and/or drug abusers;
6. Subjects with any pre-operative findings identified by the surgeon that may preclude conduct of the study procedure.

   Intra-operative:
7. Subjects with any intra-operative findings identified by the surgeon that may preclude the use of study product;
8. Subject with TBS in an actively infected field [Class III Contaminated or Class IV Dirty or Infected (see Appendix 2 in in Section 15.2)];
9. TBS is on arteries or veins where application of SURGICEL Powder would present a risk of introducing the study product into an open blood vessel;
10. Major arterial or venous bleeding or major defects in arteries and veins;
11. TBS where silver nitrate or any other escharotic chemicals have been applied;
12. TBS is in, around, or in proximity to foramina in bone, or areas of bony confine, the spinal cord, or optic nerve and chiasm;
13. TBS in urological procedures where plugging (blocking) of the urethra, ureter or a catheter is possible by the study product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2020-06-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Belgium (2):
  - Ziekenhuis Oost Limburg, Genk
  - Universitair Ziekenhuis Gent, Ghent
- United Kingdom (6):
  - NHS Lothian (Western General Hospital), Edinburgh, Lothian
  - Cambridge University Hospitals NHS Trust (Addenbrooke's Hospital), Cambridge
  - Golden Jubilee National Hospital, Clydebank
  - Leeds Teaching Hospitals NHS Trust (St James's University Hospital), Leeds
  - Newcastle upon Tyne NHS Foundation Trust (Freeman Hospital), Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottingham

REFERENCES:
- [Derived] Al-Attar N, de Jonge E, Kocharian R, Ilie B, Barnett E, Berrevoet F. Safety and Hemostatic Effectiveness of SURGICEL(R) Powder in Mild and Moderate Intraoperative Bleeding. Clin Appl Thromb Hemost. 2023 Jan-Dec;29:10760296231190376. doi: 10.1177/10760296231190376. PMID 37501509

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened up to 21 days prior to surgery and attended a baseline visit within 24 hours of surgery. Both visits took place at a clinic within the hospital where surgery also took place. Subjects were followed until hospital discharge and requested to attend a visit at 30 (+14) days post surgery and at 6 months (+/- 30 days) either at the hospital or via telephone.
Pre-assignment Details: Subjects required to meet pre-defined inclusion/exclusion criteria prior to receiving study product. Subjects required to have an appropriate mild or moderate target bleeding site (TBS) identified intra-operatively. Subjects excluded if the TBS was where silver nitrate or any other escharotic chemicals were applied, was in, around, or in proximity to foramina in bone, areas of bony confine or where plugging of the urethra, ureter or a catheter was possible by study product.
Groups:
- SURGICEL Powder: Absorbable Haemostatic Powder (Oxidized Regenerated Cellulose)
Period: Overall Study
Arm/Group | SURGICEL Powder
Started | 103
Completed | 101
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | SURGICEL Powder
Number analyzed (Participants) | 103
Age, Continuous [Median (Full Range); unit: Years]
  Age at Consent | 64.0 [33.0 to 88.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 52
Race/Ethnicity, Customized [Number; unit: Participants]
  Race : White | 93
  Race : Asian | 2
  Race : Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Haemostatic Success at 5 Minutes
Description: Proportion of subjects achieving haemostatic success at 5 minutes following application of SURGICEL Powder with no rebleeding requiring additional treatment at the Target Bleeding Site (TBS) any time prior to initiation of final fascial closure
Time Frame: From application of SURGICEL Powder to 5 minutes after application
Population: Intent to Treat (All subjects for whom TBS was identified)
Measure: Count of Participants; unit: Participants
Arm/Group | SURGICEL Powder
Number analyzed (Participants) | 103
Participants | 90
Statistical Analysis 1: Comparison: SURGICEL Powder; Test type: Other — Confidence Interval; percentage of sucesses = 87.4, 95% CI 2-sided [79.4 to 93.1]

2. Secondary Outcome: Haemostatic Success at 3 Minutes
Description: Proportion of subjects achieving haemostatic success at 3 minutes following application of SURGICEL Powder with no rebleeding requiring additional treatment at the TBS any time prior to initiation of final fascial closure
Time Frame: From application of SURGICEL Powder to 3 minutes after application
Measure: Count of Participants; unit: Participants
Arm/Group | SURGICEL Powder
Number analyzed (Participants) | 103
Participants | 80
Statistical Analysis 1: Comparison: SURGICEL Powder; Test type: Other — Confidence Interval; Percentage of Successes = 77.7, 95% CI 2-sided [68.4 to 85.3]

3. Secondary Outcome: Haemostatic Success at 10 Minutes
Description: Proportion of subjects achieving haemostatic success at 10 minutes following the application of SURGICEL Powder with no rebleeding that requires additional treatment at the TBS any time prior to initiation of final fascial closure
Time Frame: From application of SURGICEL Powder to 10 minutes after application
Measure: Count of Participants; unit: Participants
Arm/Group | SURGICEL Powder
Number analyzed (Participants) | 103
Participants | 95
Statistical Analysis 1: Comparison: SURGICEL Powder; Test type: Other — Confidence Interval; Percentage of Successes = 92.2, 95% CI 2-sided [85.3 to 96.6]

4. Other Pre Specified Outcome: Number of Participants Experiencing a Thromboembolic Event
Description: Number of participants experiencing a thromboembolic event that was assessed as having either an unlikely, possible, probable or causal relationship to the study treatment
Time Frame: From application of SURGICEL Powder to 30 day follow-up visit
Measure: Count of Participants; unit: Participants
Arm/Group | SURGICEL Powder
Number analyzed (Participants) | 103
Participants | 0

5. Other Pre Specified Outcome: Number of Participants With Post-operative Re-bleeding
Description: Number of participants of post-operative re-bleeding that was assessed as having either an unlikely, possible, probable or causal relationship to the TBS and requiring medical/surgical intervention
Time Frame: From initiation of final fascial closure to the 30-day follow up visit
Measure: Count of Participants; unit: Participants
Arm/Group | SURGICEL Powder
Number analyzed (Participants) | 103
Participants | 0

6. Other Pre Specified Outcome: Number of Participants Experiencing a Serious Adverse Events Requiring Surgical Intervention and Related to SURGICEL Powder
Description: Number of participants experiencing a serious adverse event requiring surgical intervention and assessed as having either an unlikely, possible, probable or causal relationship to the study treatment
Time Frame: From time of SURGICEL Powder application to 6-month follow up visit
Measure: Count of Participants; unit: Participants
Arm/Group | SURGICEL Powder
Number analyzed (Participants) | 103
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time product applied to TBS and up to 30 (+14) day follow-up visit. From initiation of final fascial closure to 6-month follow-up visit, SAEs requiring surgical intervention and assessed as having either an unlikely, possible, probable or causal relationship to the study treatment were recorded.
Description: For this study, an AE is an untoward medical occurrence (sign, symptom or disease) in a subject and which does not necessarily have a causal relationship with the study medical device. An untoward medical occurrence includes any new, undesirable medical experience or worsening of a pre-existing condition.
Arm/Group | SURGICEL Powder
All-Cause Mortality (participants affected / at risk) | 2/103
Serious Adverse Events (participants affected / at risk) | 24/103
Other Adverse Events (participants affected / at risk) | 63/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SURGICEL Powder (N=103)
Heart rate irregular (Investigations) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
Pancreatic fistula (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Device related sepsis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemodynamic instability (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Death (General disorders) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SURGICEL Powder (N=103)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Iron Deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Thromobocytosis (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Pericardial effusion (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 6 (6)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 6 (6)
Impaired gastric emptying (Gastrointestinal disorders) | 3 (3)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 22 (23)
Obstruction gastric (Gastrointestinal disorders) | 1 (1)
Steatorrhoea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 11 (12)
Chest pain (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Inflammation (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 4 (5)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (2)
Bacterial infection (Infections and infestations) | 1 (1)
Biliary tract infection bacterial (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Escherichia infection (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5)
Wound infection (Infections and infestations) | 5 (5)
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Gastroparesis postoperative (Injury, poisoning and procedural complications) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 9 (9)
Wound dehiscence (Injury, poisoning and procedural complications) | 3 (3)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1)
Bile culture positive (Investigations) | 1 (1)
Blood lactic acid increased (Investigations) | 2 (2)
Blood magnesium decreased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 2 (2)
Body temperature increased (Investigations) | 1 (1)
Haematocrit decreased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Prothrombin time prolonged (Investigations) | 1 (1)
Red blood cell count decreased (Investigations) | 1 (1)
Urine output decreased (Investigations) | 3 (3)
Weight decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 2 (2)
Anorexia nervosa (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pityriasis rubra pilaris (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 5 (5)
Hypotension (Vascular disorders) | 7 (7)
Thrombophlebitis superficial (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication based on results shall not be made before the first multi-centre publication.

Trust and/or Investigator may prepare data derived from the Clinical Investigation for publication. Sponsor to be given at least 60 days for review. During review period, Sponsor is entitled to request publication be delayed for up to 6 months from date of first submission to Sponsor to enable Sponsor to take steps to protect its proprietary information and/or Intellectual Property Rights and Know How.

DOCUMENTS (2):
  • Study Protocol (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT03762200/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT03762200/SAP_001.pdf